CLINICAL TRIAL: NCT06735872
Title: Effects of Non-invasive Ventilation and High-flow Oxygen Therapy on the Lung in Hypoxemic Chest Trauma Patients, a Descriptive Experimental CT Scan Study
Brief Title: Effects of Non-invasive Ventilation Therapies on the Lung in Hypoxemic Chest Trauma Patients
Acronym: VentiChest
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL24_1116
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Lung Trauma; Lung Contusion
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: The study is experimental, descriptive, prospective and monocentric. The design is with two parallel groups where each patient is his own control. That's why there is no control group. There are two groups: one receiving ten minutes of non invasive ventilation and the other one receiving ten minutes of high flow oxygen therapy. After the treatment, each participant will have an additional chest CT to determine lung volumes.
  To determine which group the participant is in, we use a randomisation without stratification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non invasive ventilation (Experimental): This group will receive a unique 10-minute session of non invasive ventilation with standard parameters directly on the CT table. The treatment will be delivered via a naso-buccal mask.
  Interventions: Procedure: Non invasive ventilation (NIV)
- High flow oxygen therapy (Experimental): This group will receive a unique 10-minute session of high flow oxygen directly on the CT table. The treatment will be delivered via a nasal cannula
  Interventions: Procedure: High flow oxygen therapy (HFO)

INTERVENTIONS:
Procedure: Non invasive ventilation (NIV) — This group will receive a unique 10-minute session of non invasive ventilation with standard parameters directly on the CT table. The treatment will be delivered via a naso-buccal mask.
  Prior to treatment, each participant will have a planned standard care chest CT.
  During the session, a senior intensivist watching for participant's comfort and safety.
  Arms: Non invasive ventilation
Procedure: High flow oxygen therapy (HFO) — This group will receive a unique 10-minute session of high flow oxygen directly on the CT table. The treatment will be delivered via a nasal cannula.
  Prior to treatment, each participant will have a planned standard care chest CT.
  During the session, a senior intensivist watching for participant's comfort and safety.
  Arms: High flow oxygen therapy

SUMMARY:
Chest trauma is common in traumatology. Its management is based on ventilatory therapies, among which non-invasive ventilation (NIV) is commonly used. Some studies have shown the benefit of this therapy in hypoxemic patients, avoiding intubation, reducing length of stay and healthcare costs, and even reducing mortality. However, these studies are old and underpowered. High flow oxygen therapy (HFO), which is frequently used in everyday practice, has only one study in chest trauma.

There is still a lack of data to really understand the effects of these techniques on the injured lung after trauma. Therefore, the investigators want to do a NIV or HFO session and directly assess the effects on participants' lungs by doing a CT at the end of the session.

This is a procedure carried out within five days of the initial trauma and consists of either a 10-minute session of non-invasive ventilation or a 10-minute session of high-flow oxygen therapy, depending on which arm the participant is allocated to.

Two chest CTs will be performed: the first as part of usual care before the non-invasive ventilation session or high flow oxygen therapy session, and the second immediately after the 10-minute session.

The investigator's objective is to demonstrate an improvement in lung recruitment with NIV or HFO using CT imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Chest trauma < 5 days
* At least 3 ribs fracture on initial CT-scan
* Need of oxygen moderated to maintain monitoring oxygen saturation Sp02 > 92% or partial pressure of arterial oxygen Pa02/ Fraction of inspired oxygen FiO2 > 200
* Intensive Care Unit admission
* Need a chest CT control during the five first days after the trauma

Exclusion Criteria:

* Patient intubated or with respiratory failure : measured or estimated Pa02/FiO2 < 200 or indication for intubation (several with respiratory rate > 35/min, abundant tracheal secretions, significant increase in work of accessory respiratory muscles on inspiration, signs of respiratory exhaustion on arterial blood gas with The potential of Hydrogen pH < 7,3 or PaCO2 > 50 mmHg, severe hypoxemia with PaO2/FiO2 ratio < 100 or desaturation < 88% for more than 5 minutes)

  * Inability to maintain 10 seconds of apnoea required for scan acquisition
  * Patient treated with ventilatory support by NIV or HFO in the 12 hours prior the investigation
  * Uncontrolled circulatory failure with need for introduction of Noradrenaline > 0,15 ug/kg/min
  * Uncontrolled neurological failure with Glasgow Coma Scale (CGS < 15
  * Unstable facial trauma or with pneumocephalus or basilar skull trauma
  * Large, undrained pneumothorax with lateral separation at the level of the hilum > 2 cm and extensive throughout the axillary line
  * Patients with identified cognitive impairment
  * Persons deprived of liberty, persons under protective measures
  * Persons not affiliated to a social security insurance
  * Current pregnancy or breastfeeding
  * Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2027-04-22 (Estimated); Study Completion 2027-04-22 (Estimated)

PRIMARY OUTCOMES:
lung volume | At day 0
  The primary outcome is evaluated by a quantitative method to compare lung volumes before and after ventilations sessions. The aim is to measure pulmonary recruitment which corresponds to the lung volume reaerated by ventilatory techniques (NIV and HFO), meaning the difference between the non-aerated lung volume between after and before the intervention. Thus, recruitment includes the partial or total re-aeration of lung areas initially not aerated before the intervention.
  The senior radiologist determine the non aerated volumes on mm3 thanks to a dedicated software. We will use a semi-automatic segmentation can be carried out quickly and reproducibly.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Edouard Herriot, Lyon, Rhône, France